CLINICAL TRIAL: NCT02769767
Title: Association of Polymorphisms of the Interleukin-7 Receptor-α (IL-7R), Glypican 5 (GPC5), Interleukin-2 Receptor-α (IL2-RA) , Human Leukocyte Antigen Class II Beta Chain (HLA-DRB1) Genes and Treatment Response in Multiple Sclerosis (MS).
Brief Title: Polymorphisms of Interleukins, Glypican, and Human Leukocyte Antigen Genes and Treatment Response in Multiple Sclerosis.
Acronym: WESTEMDRB1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Jalisciense de Cancerologia (Other Government)
Collaborators: Instituto Mexicano del Seguro Social (Other Government); University of Guadalajara (Other)
Responsible Party: Principal Investigator, Jose Alfonso Cruz-Ramos, Research Coordinator, Instituto Jalisciense de Cancerologia
Other Study IDs: EM-1
Record Dates: First submitted 2016-04-25; First posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Glypicans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Total blood for posterior extraction of DNA.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Cases: Subjects with Relapsing-Remitting Multiple Sclerosis. Polymorphisms frequencies of Interleukins, Glypican, and Human Leukocyte Antigen Genes are determined.
  Interventions: Genetic: Polymorphism of Interleukins, Glypican, and Human Leukocyte Antigen Genes.
- Controls: Healthy subjects. Polymorphisms frequencies of Interleukins, Glypican, and Human Leukocyte Antigen Genes are determined.
  Interventions: Genetic: Polymorphism of Interleukins, Glypican, and Human Leukocyte Antigen Genes.
- Responders: Subjects with MS treated for at least two years that have less than one relapse per year or who had an increase of <1.5 points on the Expanded Disability Status Scale (EDSS) (if baseline EDSS was 0) or no increase in EDSS (baseline EDSS ≥1). Polymorphisms frequencies of Interleukins, Glypican, and Human Leukocyte Antigen Genes are determined.
  Interventions: Genetic: Polymorphism of Interleukins, Glypican, and Human Leukocyte Antigen Genes.
- No responders: Subjects with MS that have more than one relapse per year treated for at least two years, and who had ≥1 relapse(s) or an increase of 1.5 points on the EDSS (if baseline EDSS was 0) or an increase of ≥0.5 points (baseline EDSS ≥1). Polymorphisms frequencies of Interleukins, Glypican, and Human Leukocyte Antigen Genes are determined.
  Interventions: Genetic: Polymorphism of Interleukins, Glypican, and Human Leukocyte Antigen Genes.

INTERVENTIONS:
Genetic: Polymorphism of Interleukins, Glypican, and Human Leukocyte Antigen Genes. — The frequencies of the polymorphic variants in subjects with MS and healthy subjects were evaluated. Also in subjects with MS, the response to treatment with the number of relapses and EDSS was assessed; to compare the allele frequencies of SNPs of Interleukins, Glypican, and Human Leukocyte Antigen Genes, between responders and no responders MS patients.

SUMMARY:
HLA-DRB1 * Gene and some genes involved in inflammation and immunity (IL-7R, GPC5, CTSS) have been linked to risk of MS and the response to treatment with immunomodulators. This research aims to estimate the risk that confers some variations in the sequence of these genes.

DETAILED DESCRIPTION:
Genes HLA-DRB1 * and some genes involved in inflammation and immunity have been linked to risk of MS and the response to treatment with immunomodulators.

The HLA-DRB1 * genes have been associated with risk and response to treatment in MS in multiple studies; however, other genes have been controversial. This research aims to estimate the risk for MS that confers some variations in the sequence of IL-7R, GPC5, CTSS, HLA-DRB1 genes. Furthermore, it seeks to determine whether these gene variants (polymorphisms) are associated with treatment response to immunomodulators.

Subjects with MS and healthy subjects will be taken to assess the risk for MS. Besides the investigators obtain the medical history of relapse to assess response to treatment in accordance with Expanded Disability Status Scale (EDSS) and relapses.

ELIGIBILITY:
Inclusion Criteria for Cases:

* Subjects with multiple sclerosis
* 18 and over
* EDSS less than 5
* Signed informed consent

Inclusion Criteria for Controls:

* Healthy subjects
* 18 and over
* Signed informed consent

Exclusion Criteria for Cases:

* Mental retardation
* Withdrawal of consent
* No immunomodulatory treatment

Exclusion Criteria for Controls:

* Mental retardation
* Withdrawal of consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with multiple sclerosis and healthy subjects were studied. In subjects with multiple sclerosis, the number of relapses and EDSS was evaluated for two years.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Treatment response evaluated by relapses per year, evaluated during two years after recruitment. | Two Years
  Treatment response evaluated by relapses per year during two years after recruitment. The relapses are defined by any neurological sign or symptom that happens at least 30 days after any previous neurological deterioration episode began.
Treatment response evaluated by Expanded Disability Status Scale (EDSS) during two years after recruitment. | Two Years
  Treatment response evaluated by Expanded Disability Status Scale (EDSS) during two years after recruitment.
  The EDSS scale ranges from 0 to 10; the increments are in 0.5. Scoring is based on an examination by a neurologist about the level of disability.

SECONDARY OUTCOMES:
Multiple Sclerosis Risk Conferred by Single Nucleotide Polymorphisms (SNPs) of Interleukins, Glypican, and Human Leukocyte Antigen Genes. | One Year
  The risk conferred by SNPs of Interleukins, Glypican, and Human Leukocyte Antigen Genes: calculated by odds ratio when the allele frequencies of SNPs cases are compared with the allele frequencies of SNPs in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: JOSE A. CRUZ RAMOS, PhD, Principal Investigator — Instituto Jalisciense de Cancerología
Locations (1):
- Instituto Jalisciense de Cancerología, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided